CLINICAL TRIAL: NCT05730478
Title: Comparison Between Anterior Segment Optical Coherence Tomography and Ultrasound Bio Microscopy Parameters in Glaucoma Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Adel Omar, Resident doctor at ophthalmology department in sohag teaching hospital, Sohag University
Other Study IDs: MAOmar
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma Eye

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ASOCT and UBM parameters Comparison: comparison between ASOCT and UBM parameters in glaucoma ASSESMENT
  Interventions: Device: ASOCT&UBM; Drug: Glaucoma therapy

INTERVENTIONS:
Device: ASOCT&UBM — glaucoma assesment by ASOCT &UBM
Drug: Glaucoma therapy — ASOCT and UBM parameters Comparison
Drug: Glaucoma therapy — Comparison
  Other Names: ASOCT

SUMMARY:
Study aiming to compare between anterior segment Optical Coherence Tomography and Ultrasound BioMicroscopy In Glaucoma aSSESMENT

DETAILED DESCRIPTION:
Glaucoma is comprised of a group of optic neuropathies that share certain biological and clinical characteristics including progressive loss of the RGCs that causes specific, irreversible changes to the optic disc and visual field Visualization of the anterior chamber (AC) angle is a critical step in the diagnosis of glaucoma, especially angle-closure variants. .

UBM has been used in imaging and quantitative evaluation of anterior ocular segments since the 1990s. It allows in vivo observation of the anatomy and pathology of the anterior segments, from the conjunctiva and cornea to the iris and basal vitreous body, which provides significant information on glaucoma, cysts, neoplasms, trauma and foreign bodies. UBM also provides biometric information of anterior segment structures, such as anterior chamber (AC) depth, anterior chamber angle (ACA), and iris thickness. UBM provides more detailed information compared to slit-lamp, gonioscopy or B-scan examinations for diagnosis and follow-up of PAC eyes.In some cases UBM elucidates the mechanism of elevated intraocular pressure by showing the relationship between the peripheral iris and the trabecular meshwork. It can be used to study the causes of secondary glaucoma, for example, the pigment dispersion syndrome, lens-induced glaucoma, ciliary block, cysts, and solid tumors of the anterior segment. It can also assess the effects of various interventions such as laser iridotomy, trabeculectomy, and non-penetrating drainage surgery. Precise quantitative evaluation of the anterior chamber angle structures can help in diagnosis and management of various pathologies related to glaucoma . Optical coherence tomography (OCT) is a widely used non-invasive fundus imaging technique. Since the first application of OCT in the cornea in 2002], anterior segment-optical coherence tomography (AS-OCT) has developed rapidly. There are two major OCT platforms on the market: time domain-optical coherence tomography (TD-OCT) and spectral (or Fourier) domain-optical coherence tomography (SD/FD-OCT) . With a higher imaging resolution than UBM, AS-OCT makes it easier for the operator and software to identify ACA structures. such as: the scleral spur (SS), iris surface, Schwalbe's line, even trabecular meshwork (TM), and Schlemm's canal. This provides more precise analysis of the angle opening distance (AOD) from the SS, ACA, trabecular iris angle (TIA), and trabecular iris space area (TISA)

ELIGIBILITY:
Inclusion Criteria:

* Patients with open and angle closure glaucoma. Male and female patients were included. Patient age: more than18 years old

Exclusion Criteria:

Previous glaucoma surgery. Previous cataract surgery. Media opacity. Associated ocular or intra ocular inflammation. Associated corneal pathology.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: comparison between anterior segment optical coherence tomography and ultrasound biomicroscopy parameters in glaucoma assesment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
comparison between Anterior Segment Optical Coherence Tomography And ltrasound Biomicroscopy Parameters In Glaucoma Assesment | 1 year
  . UBM provides biometric information of anterior segment structures, such as anterior chamber (AC) depth, anterior chamber angle (ACA), and iris thickness. UBM provides more detailed information compared to slit-lamp, gonioscopy or B-scan examinations for diagnosis and follow-up of PAC eyes. It can be used to study the causes of secondary glaucoma. Precise quantitative evaluation of the anterior chamber angle structures can help in diagnosis and management of various pathologies related to glaucoma .
  anterior segment-optical coherence tomography (AS-OCT) has developed rapidly. With a higher imaging resolution than UBM, AS-OCT makes it easier for the operator and software to identify ACA structures. such as: the scleral spur (SS), iris surface, Schwalbe's line, even trabecular meshwork , and Schlemm's canal. This provides more precise analysis of the angle opening distance from the SS, ACA, trabecular iris angle , and trabecular iris space area

CONTACTS AND LOCATIONS:
Overall Officials: Osama Ali, professor, Study Director — Sohag University; Islam Saad, Assistant, Study Director — Sohag University; Mohamed Ezz, lecturer, Study Chair — Sohag University
Locations (1):
- Marwa Adel,, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casson RJ, Chidlow G, Wood JP, Crowston JG, Goldberg I. Definition of glaucoma: clinical and experimental concepts. Clin Exp Ophthalmol. 2012 May-Jun;40(4):341-9. doi: 10.1111/j.1442-9071.2012.02773.x. Epub 2012 Apr 5. PMID 22356435
- [Background] Barkana Y, Dorairaj SK, Gerber Y, Liebmann JM, Ritch R. Agreement between gonioscopy and ultrasound biomicroscopy in detecting iridotrabecular apposition. Arch Ophthalmol. 2007 Oct;125(10):1331-5. doi: 10.1001/archopht.125.10.1331. PMID 17923539
- [Background] Dada T, Mohan S, Sihota R, Gupta R, Gupta V, Pandey RM. Comparison of ultrasound biomicroscopic parameters after laser iridotomy in eyes with primary angle closure and primary angle closure glaucoma. Eye (Lond). 2007 Jul;21(7):956-61. doi: 10.1038/sj.eye.6702360. Epub 2006 May 5. PMID 16680106
- [Background] Wirbelauer C, Scholz C, Haberle H, Laqua H, Pham DT. Corneal optical coherence tomography before and after phototherapeutic keratectomy for recurrent epithelial erosions(2). J Cataract Refract Surg. 2002 Sep;28(9):1629-35. doi: 10.1016/s0886-3350(02)01366-4. PMID 12231324
- [Background] Reinstein DZ, Gobbe M, Archer TJ. Anterior segment biometry: a study and review of resolution and repeatability data. J Refract Surg. 2012 Jul;28(7):509-20. doi: 10.3928/1081597X-20120620-02. PMID 22767168
- [Background] Sharma R, Sharma A, Arora T, Sharma S, Sobti A, Jha B, Chaturvedi N, Dada T. Application of anterior segment optical coherence tomography in glaucoma. Surv Ophthalmol. 2014 May-Jun;59(3):311-27. doi: 10.1016/j.survophthal.2013.06.005. Epub 2013 Oct 15. PMID 24138894
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22356435/